CLINICAL TRIAL: NCT04664842
Title: Effect of Diaphragmatic Stretch Technique and Breathing Exercise Intervention in Patients With Chronic Neck Pain
Brief Title: Effects of Manual Therapy and Exercise Training of Diaphragm in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, YI-JU TSAI, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCKU_Diaphragm
Record Dates: First submitted 2020-09-04; First posted 2020-12-11 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Chronic Neck Pain
Keywords: Ultrasonography; Diaphragm; Breathing exercise; Breathing dysfunction
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Manual Therapy Group (Experimental)
  Interventions: Other: Diaphragmatic Stretch Technique
- Manual Control Group (Sham Comparator)
  Interventions: Other: Diaphragmatic Stretch Technique
- Breathing Training Group (Experimental)
  Interventions: Other: Breathing Exercise Training
- General Exercise Control Group (Sham Comparator)
  Interventions: Other: Breathing Exercise Training
- Manual Therapy Combined Breathing Training Group (Experimental)
  Interventions: Other: Diaphragmatic Stretch Technique; Other: Breathing Exercise Training

INTERVENTIONS:
Other: Diaphragmatic Stretch Technique — Diaphragmatic stretch technique is an intervention intended to indirectly stretch the diaphragmatic muscle fibers. This will help to decease tension generated by trigger points, normalizing muscle ﬁber length, and improve muscle contraction.
  Arms: Manual Control Group; Manual Therapy Combined Breathing Training Group; Manual Therapy Group
Other: Breathing Exercise Training — During diaphragmatic or abdominal breathing training, inhalation will caused diaphragm contract downwards, inflating the lungs. This filling of the lungs pushes the abdominal organs down leading to expansion of the abdomen. Subjects are required to do few repetitions during the intervention.
  Arms: Breathing Training Group; General Exercise Control Group; Manual Therapy Combined Breathing Training Group

SUMMARY:
Chronic neck pain is a commonly reported problem and often associated with functional disability. Studies showed that patients with chronic neck pain compensated with changes in breathing pattern. Primary functions of the diaphragm includes as the main respiratory muscle and contributing to the postural stability and spinal control. Diaphragm is located between the thorax and abdomen and has extensive and complex fascial connections to surrounding organs, muscles, and skeletons. Few studies showed that applying diaphragmatic manual techniques and breathing exercise training help to improve functions in patients with low back pain. However, how does the interventions directly influence on patients with chronic neck pain is still unclear. In this study, we make a hypothesis that diaphragmatic stretch technique and breathing exercise training help to reduce pain and improve functions in patients with chronic neck pain.

DETAILED DESCRIPTION:
Chronic neck pain is a serious health problem with low quality of life, disability and economical burdens. Studies have found that nearly 83% of chronic neck pain patients had changes in breathing patterns. Compensated breathing pattern by using the neck-accessory respiratory muscles may result in excessive muscle strains and over-activations, which may also contribute to develop chronic neck pain. The diaphragm is the most important respiratory muscle which attached to the ribs and spine, and thus has an influence on spinal stability. Few studies have showed that diaphragm releasing and breathing training can reduce pain and improve flexibility of posterior chain muscles, spinal range of motions, and ribcage excursions in asymptomatic adults and patients with low back pain. However, the effects in patients with chronic neck pain has not bee determined. Therefore, there are two main purpose of this study. First, to determine the relationships among diaphragm mobility, neck pain and dysfunction, and respiratory in patients with chronic neck pain. Second, to investigate the effects of diaphragm releasing, breathing training, or combined intervention on pain and disability in patients with chronic neck pain. It is expected to recruit 150 patients with chronic neck pain and 30 healthy volunteers. Patients with chronic neck pain will be randomly assigned to (1) manual therapy group (2) manual control group (3) breathing training group (4) general exercise control group (5) manual therapy combined breathing training group. Each participant will receive a specific intervention program depending on their group allocation. All participants will receive two evaluation sessions before and after the intervention including ultrasonography, cervical and thoracic function, respiratory functions, and autonomic balance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic or recurrent neck pain from upper cervical to T1 area
* Condition last for 3 months and above

Exclusion Criteria:

* Acute neck pain
* Previous neck, shoulder or thoracic surgery
* Neurological disease
* Cardiopulmonary disease（Eg. Chronic obstructive pulmonary disease (COPD), pulmonary tuberculosis (TB), asthma, chronic bronchitis, pulmonary emphysema）
* Smoking
* Pregnancy
* Tumour
* Psychological disease
* Neuromuscular disease
* Back pain
* Anaemia or Diabetes
* Neck rehabilitation for past 12 month
* Scoliosis or other diseases that cause spine and chest deformity
* BMI > 30

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Change from baseline pain intensity up to 2 weeks
  Visual Analog Scale: Minimum value = 0 (Best outcome); Maximum value = 10 (Worst Outcome)

SECONDARY OUTCOMES:
Functional Disability | Change from baseline functional disability up to 2 weeks
  Neck disability index - Questionnaire

OTHER OUTCOMES:
Neck and Thoracic ROM | Change from baseline neck and thoracic ROM up to 2 weeks
  Dual inclinometer
Neck Muscle Endurance | Change from baseline neck muscle endurance up to 2 weeks
  Electromyography: EMG amplitude (root mean square, RMS) and frequency (median frequency, MF) on neck muscle
Neck Muscle Strength | Change from baseline neck muscle strength up to 2 weeks
  Micro FET2
Chest Mobility | Change from baseline check mobility up to 2 weeks
  Tape ruler
Diaphragmatic Changes | Change from baseline diaphragmatic chages up to 2 weeks
  Diaphragmatic thickness, mobility and strength using ultrasonography (M mode, B mode)
Maximal Inspiratory Pressure (MIP), Maximal Expiratory Pressure (MEP) | Change from baseline MIP and MEP up to 2 weeks
  Gas pressure gauge
Lung Function | Change from baseline lung function up to 2 weeks
  Forced Vital Capacity (FVC), Forced Expiratory volume in one second (FEV1) using Spirometer
Heart Rate Variability | Change from baseline heart rate variability up to 2 weeks
  Hand-held Electrocardiogram (CheckMyHeart Plus)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, East District, Taiwan

REFERENCES:
- [Derived] Cheng KC, Hii EYX, Lin YN, Kuo YL, Tsai YJ. Effects of manual diaphragm release on pain, disability and diaphragm function in patients with chronic neck pain: a pilot randomized controlled trial. BMC Complement Med Ther. 2025 Oct 1;25(1):349. doi: 10.1186/s12906-025-05090-8. PMID 41034882